CLINICAL TRIAL: NCT06202508
Title: Fetal Death in Utero in the Internship Experience of Midwifery Students : an Unavoidable Experience?
Acronym: MFU
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8335
Record Dates: First submitted 2022-12-14; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Fetal Death in Utero
Keywords: Fetal death in utero
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal death in utero and the psychological and professional impact it could have on the midwifery student in training. Fetal death in utero corresponds to the spontaneous cessation of cardiac activity, from 14 weeks of amenorrhea.

For a large proportion of midwifery students, fetal death in utero is a situation encountered in the field. Despite the theoretical courses, a student does not expect to encounter this type of situation during the internship: it is delicate for both the supervising caregivers and the student. The purpose of this study is to demonstrate the impact that this situation could have on the midwifery student, both psychologically and in terms of their professional project.

DETAILED DESCRIPTION:
The aim of the research is to highlight the psychological and professional impact of in utero fetal death among midwifery students in Strasbourg.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years
* Midwifery student of the Strasbourg school of medicine of 3rd year or more
* having experienced the discovery of a fetal death in utero in a birth room internship
* having participated in the follow-up of an in utero fetal death in the birth room
* Agreed to participate in the interview and did not express opposition to the reuse of their data for the purpose of this research

Exclusion Criteria:

- Subject who expressed opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Midwifery student of the Strasbourg school of medicine having experienced the discovery of a fetal death in utero in a birth room internship
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
To highlight the psychological and professional impact of in utero fetal death on Strasbourg midwifery students. | Approximately 10 months after a midwifery student was in charge of a case of fetal death in utero
  Analysis of midwifery students' experiences during their internship in Strasbourg through semi-directive interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France